CLINICAL TRIAL: NCT04518852
Title: TACE Combined With Sorafenib and PD-1 mAb in the Treatment of BCLC B/C Hepatocellular Carcinoma: Single Arm, Single Center, Open Label Study
Brief Title: TACE, Sorafenib and PD-1 Monoclonal Antibody in the Treatment of HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Guohui Xu, Sichuan Cancer Hospital and Research Institute, Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GXu
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma; Liver Neoplasms; Digestive System Neoplasms; Sorafenib; Molecular Mechanisms of Pharmacological Action; Liver Diseases; Antineoplastic Agents; Protein Kinase Inhibitors
Keywords: Hepatic Artery Embolism; Angiogenesis; Immune Suppression
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Digestive System Neoplasms; Liver Diseases | interventions — Sorafenib

STUDY DESIGN:
Intervention Model Description: This study focuses on the in-operable, BCLC-B/C stage HCC patients. The participants will receive the combined treatment of local therapy (TACE) , anti-angiogenic therapy (sorafenib), and immunotherapy (PD-1 monoclonal antibody)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): The participants will receive the combined treatment of local therapy (TACE, oxaliplatin and epirubicin), anti-angiogenic therapy (sorafenib), and immunotherapy (PD-1 monoclonal antibody)
  Interventions: Combination Product: TACE combined with sorafenib and PD-1 mAb

INTERVENTIONS:
Combination Product: TACE combined with sorafenib and PD-1 mAb — the combination of local therapy (TACE), anti-angiogenic therapy (sorafenib), and immunotherapy (PD-1 monoclonal antibody)

SUMMARY:
Hepatocellular carcinoma (HCC) is the fourth most common cause of cancer-related death that ranks sixth in terms of incident cases, with an overall 5 years survival of 18%. Despite a significant improvement in treatment strategy, the overall survival of HCC remains low due to high recurrence, progressive liver dysfunction and the high fatality of the disease. Surgical resection has been applied in a number of patients; however, surgery has been associated with a high incidence of recurrence (approximately 70% within 5 years). TACE is generally applied on intermediate-stage HCC. However, TACE is not satisfied with improving overall survival. Therefore, there is an urgent need for effective treatment for these patients.

At present, the overall objective response rate (ORR) of single or sequential therapy is not satisfied, and the over survival (OS) improvement is not ideal. Therefore, combined therapy maybe the good choice for patients with advanced HCC.

This study focuses on the in-operable, BCLC-B/C HCC patients. Through the combination of local therapy (TACE), anti-angiogenic therapy (Sorafenib), and immunotherapy (PD-1 monoclonal antibody), it is expected to change the tumor microenvironment, restore the immune response, strengthen the anti-tumor effect of various treatments, and improve the therapeutic efficacy in patients with BCLC-B/C HCC.

DETAILED DESCRIPTION:
This study is a single arm, single center, open label study. It is estimated that 60 patients with BCLC-B/C HCC who can not receive radical resection will be enrolled.

The trial period of subjects includes screening period, treatment period and follow-up period.

The drug treatment was 200 mg of PD-1 monoclonal antibody, intravenous infusion on the first day, every 21 days as a treatment cycle; mesylate sorafenib, 400 mg, oral twice a day, continuous oral; TACE, the lipiodol + blank microspheres and oxaliplatin (100 mg) + epirubicin (50 mg) were injected into the hepatic artery by routine procedure, repeated every 4-6 weeks, and administered for according to the physician in charge, TACE treatment cycles. Treatment continues until the disease progresses, intolerable toxicity occurs, new anti-tumor treatment is started, informed consent is withdrawn, follow-up is lost, death occurs or treatment termination is required。 Screening will be performed between days - 21 and - 4. Informed consent was signed up to 4 weeks prior to the first day of cycle 1 before any screening procedure or evaluation was performed and the trial was fully explained to each subject.

Baseline evaluation results must be collected prior to the first trial drug administration (day 1 of cycle 1). Baseline assessments may be performed between days - 3 and - 1 or on day 1 of cycle 1. If performed within 3 days before the first day of cycle 1, the screening results can be used as baseline results.

The tumor imaging was evaluated every 4-6 weeks since the first administration, and every 12 weeks (± 7 days) after 24 weeks. If there are clinical indications for disease progression, tumor evaluation is more frequent. In the event of disease progression, unacceptable toxicity, the subject's request to discontinue the trial or the subject's withdrawal of consent, the subject will discontinue the trial treatment.

When the trial treatment is stopped, the treatment visit shall be stopped within 7 days after the treatment is stopped in order to stop the treatment examination.

After the end of the treatment period (up to 2 years), subjects who can benefit from the study drug will continue to study the treatment of the drug until disease progression, intolerable adverse reactions, withdrawal of intensive care facility (ICF), other anti-tumor treatment, loss of follow-up, death or termination of the study.

After the occurrence of a clinical event, if it is judged by the investigators that it should be attributed to the progress of the disease and it is unlikely to recover even if the patient continues to receive treatment, it can be evaluated as clinical deterioration. It is up to the investigator to discuss and decide whether to continue or stop the treatment for the subject and record in the study file.

At the end of the study, subjects who are still under study treatment can continue to receive treatment through another extended study or other forms at the discretion of the investigator if they are stable or relieved in the efficacy evaluation and can tolerate the adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or clinically confirmed hepatocellular carcinoma.
2. Age ≥ 18 years old.
3. Performance status (PS) ≤ 2 (ECOG scale).
4. Barcelona clinical liver cancer (BCLC) stage B or stage C.
5. Participants who have not received other systemic anti-tumor treatment for HCC before the first administration.
6. Patients who had not received TACE before the first administration, or who had received 0-2 times TACE but PD or SD ≥ 4 weeks.
7. According to mRECIST, there is at least one measurable lesion.
8. Child Pugh score ≤ 7.
9. Participant has sufficient organ and marrow functions.
10. Expected survival time ≥ 12 weeks.
11. For women of childbearing age or male patients whose sexual partners are women of childbearing age, effective contraceptive measures should be taken during the whole treatment period and 6 months after the last medication.
12. Sign the written informed consent, and be able to follow the visit and relevant procedures specified in the plan

Exclusion Criteria:

1. Fibrolamellar carcinoma, sarcomatoid carcinoma, cholangiocarcinoma and other components previously confirmed by histology / cytology.
2. History of hepatic encephalopathy or liver transplantation.
3. Pleural effusion, ascites and pericardial effusion with clinical symptoms requiring drainage.
4. Tumor burden≥70%, diffuse liver cancer or tumor is not suitable for mRECIST standard evaluation.
5. Received local treatment (ablation therapy), surgery resection and radiotherapy for liver cancer before the first administration.
6. Have received systemic chemotherapy, targeted therapy or immunotherapy
7. There is a significant decrease in white blood cells and platelets in peripheral blood, severe coagulation dysfunction and can not be corrected：the neutrophil<1.5×109/L, PLT<50×109/L. The INR>2.3
8. Acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV-DNA) > 10^6 copies / ml; hepatitis C virus (HCV-RNA) > 10^3 copies / ml; HBsAg and anti HCV antibody were positive at the same time.
9. There is central nervous system metastasis.
10. Bleeding of esophageal or gastric varices caused by portal hypertension occurred in the past 6 months, or severe (G3) varices were found in endoscopic examination within 3 months before the first administration, or evidence of portal hypertension (including splenomegaly found in imaging examination) was found. The researchers assessed that the risk of bleeding was high and did not receive sclerotherapy or ligation under the endoscope.
11. The previous 6-month history of arteriovenous thromboembolism, including myocardial infarction, unstable angina, cerebrovascular accident, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism. The thrombus of implanted vein port or catheter source or superficial vein is stable after routine anticoagulant treatment. Prophylactic use of low- molecular-weight heparin (e.g., enoxaparin 40 mg / day) is permitted.
12. Tumor thrombus of main portal vein, or involving superior mesenteric vein at the same time.
13. Aspirin (> 325 mg / day) or other drugs known to inhibit platelet function such as dipyridamole or clopidogrel were used for 7 consecutive days within 2 weeks before the first administration.
14. For uncontrolled hypertension, systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg after the best medical treatment, hypertension crisis or hypertension encephalopathy history.
15. Symptomatic congestive heart failure (New York Heart Association class II-IV). Symptomatic or poorly controlled arrhythmias. The corrected QT interval (QTc) for the history or screening of congenital long QT syndrome was more than 500 ms (calculated by Fridericia method).
16. Serious bleeding tendency or coagulation dysfunction, or undergoing thrombolysis.
17. In the past 6 months, there was a history of gastrointestinal perforation and / or fistula, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive enterotomy (partial colectomy or extensive enterotomy with chronic diarrhea), Crohn's disease, ulcerative colitis or long-term chronic diarrhea.
18. Previous and current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function and other lung diseases.
19. Active tuberculosis (TB), who is receiving anti TB treatment or has received anti TB treatment within one year before the first administration.
20. People with HIV infection (HIV 1 / 2 antibody positive) and known syphilis infection. Serious infection in active stage or poor clinical control.
21. Severe infection within 4 weeks before the first administration, including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia.
22. Active autoimmune diseases requiring systemic treatment (such as the use of disease alleviation drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (e.g. thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are permitted. Known history of primary immunodeficiency. Only the patients with positive autoimmune antibody need to confirm whether there is autoimmune disease according to the judgment of researchers.
23. Immunosuppressive drugs were used within 4 weeks before the first administration, excluding local glucocorticoids or systemic glucocorticoids (i.e. no more than 10 Mg / day prednisone or the equivalent dose of other glucocorticoids), allowing temporary use of glucocorticoids due to dyspnea symptoms in the treatment of asthma, chronic obstructive pulmonary disease and other diseases.
24. Receive live attenuated vaccine within 4 weeks before the first administration or during the study period.
25. Major surgical procedures (craniotomy, thoracotomy or open hand) were performed within 4 weeks before the first administration (surgery) or an unhealed wound, ulcer, or fracture.
26. Uncontrolled / uncorrectable metabolic disorder or other non- malignant organ disease or systemic disease or cancer secondary reaction, which may lead to higher medical risk and / or uncertainty of survival evaluation.
27. Known to be allergic to any PD-1 monoclonal antibody component.
28. Women of childbearing age who are unwilling or unable to use acceptable methods of contraception during the whole treatment period of this trial and within 12 weeks after the last administration of the study drug (women of childbearing age include: any women who have had menarche, and have not undergone successful artificial sterilization (hysterectomy, bilateral tubal ligation, or bilateral ovariectomy), pregnancy or lactation Women; women with positive pregnancy test results at the time of inclusion or before study drug administration; If the partner is a woman of childbearing age, the subject is a fertile male without effective contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
objective response rate (ORR) | Change from baseline tumor volume at 6 months
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit. It is the sum of the proportion of complete response (CR) and partial response(PR). That is, ORR = CR + PR
overall survival (OS) | 1 year
  the time from the beginning of treatment to death caused by any reason (the last follow-up time is for the patients who lost the visit; the end of the study is for the patients who are still alive)

SECONDARY OUTCOMES:
progression free survival (PFS) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression free survival period refers to the period from the beginning of treatment to the time when patients with cancer progress is observed or death occurs for any reason.
time to progression (TTP) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from the beginning of treatment to the objective progression of tumor
disease control rate (DCR) | 1 year
  It is the sum of the proportion of complete response (CR), partial response(PR) and stable disease(SD). That is, DCR = CR + PR + SD
duration of response | up to 48 weeks
  the time from the first evaluation of the tumor as CR or PR to the first evaluation as PD or any cause of death

OTHER OUTCOMES:
conversion rate of hepatectomy | 1 year
  The ratio of patients with locally advanced liver cancer who could not be operated on before to get radical operation through comprehensive treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China